CLINICAL TRIAL: NCT01406301
Title: Evaluate (Post Approval) the Adherence to the Prescribing Information for ARIXTRA® (Fondaparinux) in ACS Patients- Commitment of the Fondaparinux EU-RMP
Brief Title: Fondaparinux EU-RMP (Adherence)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113652; WEUSRTP2284 (Other: GSK); EPI40495 (Other: GSK)
Record Dates: First submitted 2011-07-28; First posted 2011-08-01 (Estimated); Last update posted 2015-04-27 (Estimated); Status verified 2015-04

CONDITIONS: Acute Coronary Syndrome
Keywords: prescribing information
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Fondaparinux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Patients with a discharge diagnosis of ACS (UA/NSTEMI or STEMI: Patients with a discharge diagnosis of ACS (UA/NSTEMI or STEMI)
  Interventions: Drug: fondaparinux

INTERVENTIONS:
Drug: fondaparinux — fondaparinux

SUMMARY:
Fondaparinux, a synthetic and specific factor Xa inhibitor, was granted an ACS indication by Health Canada in March 2007 and by the EMEA in September 2007. Among ACS patients, fondaparinux is indicated for the treatment of UA/NSTEMI in patients for whom urgent PCI (within 2 hours) is not indicated, and for the treatment of STEMI in patients who are managed with thrombolytics or who are initially to receive no other form of reperfusion therapy. The approved prescribing information for fondaparinux in ACS provides recommendations for use in patients undergoing PCI. The purpose of this study is to evaluate physician adherence to this prescribing information in ACS patients treated with fondaparinux and who undergo PCI. The primary endpoint is the proportion of patients with ACS treated with fondaparinux, for whom the prescribing information during PCI was followed (i.e., adjunctive anticoagulant therapy administered at the time of PCI). Measurement of the effectiveness or safety of fondaparinux use in ACS patients is not within the scope of this study.

ARIXTRA® is a trademark of the GlaxoSmithKline group of companies.

ELIGIBILITY:
Inclusion Criteria:

* Discharge diagnosis of ACS (UA/NSTEMI or STEMI)
* PCI during the hospitalization
* Anticoagulant treatment with fondaparinux

Exclusion Criteria:

* Enrollment at the time of the index hospitalization in a clinical study that could influence ACS treatment practices, specifically the in-hospital use of anticoagulation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitals with the capacity to perform cardiac catheterizations and PCIs will be identified. Sites will be further qualified based upon the expectation of an adequate number of ACS patients and the known or potential use of fondaparinux by the site. A minimum of 5 sites per country will be targeted in order to achieve a within-country representative sample. The study is planned for 7 countries in Europe and North America.
  Based on sample size estimates, approximately 32 physicians per country (6 to 7 per site) and approximately 256 patients per country (assuming an average of 8 patients per physician) will be targeted for inclusion, yielding a study total of approximately 1800 patients.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2008-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients with ACS treated with fondaparinux, for whom the prescribing information during PCI was followed (i.e., adjunctive anticoagulant therapy administered at the time of PCI) | ACS hospitalizations that occur at least one month after the availability of reimbursement for fondaparinux for the UA/NSTEMI and STEMI indications at that particular site are eligible

SECONDARY OUTCOMES:
The proportion of patients with UA/NSTEMI treated with fondaparinux, for whom the prescribing information during PCI was followed (i.e., adjunctive anticoagulant therapy administered at the time of PCI) | ACS hospitalizations that occur at least one month after the availability of reimbursement for fondaparinux for the UA/NSTEMI and STEMI indications at that particular site are eligible
The proportion of patients with STEMI treated with fondaparinux, where fondaparinux is not administered prior to or during primary PCI | ACS hospitalizations that occur at least one month after the availability of reimbursement for fondaparinux for the UA/NSTEMI and STEMI indications at that particular site are eligible
The proportion of patients with STEMI treated with fondaparinux, for whom the prescribing information during PCI was followed (i.e., adjunctive anticoagulant therapy administered at the time of PCI) | ACS hospitalizations that occur at least one month after the availability of reimbursement for fondaparinux for the UA/NSTEMI and STEMI indications at that particular site are eligible

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline